CLINICAL TRIAL: NCT05631145
Title: Morita Therapy Combined With Xingnao Kaiqiao Acupressure for Relieving Depressive Symptoms During COVID-19: A Randomized Controlled Study
Brief Title: MT Combined With XKSA for Depressive Symptoms During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Renrong Wu (Other)
Responsible Party: Sponsor-Investigator, Renrong Wu, Clinical professor, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTXKSA
Record Dates: First submitted 2022-11-28; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Depression, Anxiety
Keywords: Morita therapy; acupressure; quarantine; COVID-19; depression; anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial testing MT combined with XKSA versus MT alone.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morita therapy (MT) combined with Xingnao Kaiqiao self-administered acupressure (XKSA) (Experimental): MT combined with XKSA for 2 weeks.
  Interventions: Other: MT Combined With XKSA
- Morita therapy (MT) (Placebo Comparator): MT alone for 2 weeks
  Interventions: Other: MT

INTERVENTIONS:
Other: MT Combined With XKSA — Morita therapy (MT) comprised bed rest and light work. Xingnao Kaiqiao self-administered acupressure (XKSA) stimulates nine acupoints including Baihui, Sishenchong, Shenmen, Neiguan, Hegu, Taichong, Jianjing, Shenshu, and Yuji.
  Arms: Morita therapy (MT) combined with Xingnao Kaiqiao self-administered acupressure (XKSA)
Other: MT — Morita therapy (MT) comprised bed rest and light work.
  Arms: Morita therapy (MT)

SUMMARY:
Social isolation related mental health problems have raised many concerns during the COVID-19 outbreaks. Mental health care for people in quarantined hotels is in urgent need, but concrete program is rarely reported. Morita therapy and acupressure have been identified as effective treatments for regulating mood and sleep. The study aimed to examine whether Morita therapy (MT) combined with Xingnao Kaiqiao self-administered acupressure (XKSA) could improve depressive, anxiety symptoms and sleep quality in isolated people with depressive symptoms.

DETAILED DESCRIPTION:
The study will evaluate the efficacy and safety of Morita therapy (MT) combined with Xingnao Kaiqiao self-administered acupressure (XKSA) on ameliorating depressive, anxiety and insomnia symptoms in quarantined people with depressive symptoms by measuring changes in clinical ratings before and after all the treatments immediately. 59 participants will be randomized to receive self-administered acupressure combined with Morita therapy or Morita therapy monotherapy during the two weeks of clinical observation and quarantine in Shenzhen, China. Morita therapy (MT) comprised bed rest and light work. In the first week, the participants were instructed to stay in the room but not restrict themselves to the bed. In the second week, the therapist guided the participants to face or accept instead of deliberately eliminating negative emotions and somatic discomfort. Xingnao Kaiqiao self-administered acupressure (XKSA) protocol evolved based on the XK acupuncture techniques after consulting a Chinese medicine specialist. Other two traditional Chinese medicine experts reviewed and approved the protocol. The protocol comprised pressing nine acupoints including Baihui, Sishenchong, Shenmen, Neiguan, Hegu, Taichong, Jianjing, Shenshu, and Yuji. Changes in depressive symptoms from baseline to the end of the study will be measured by the Patient Health Questionnaire 9-item depression scale (PHQ-9). Changes in anxiety symptoms from baseline to the end of the study will be measured by the Generalized Anxiety Disorder 7-item (GAD-7). Changes in sleep quality from baseline to the end of the study will be measured by the Insomnia Severity Index (ISI).

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 65 years;
2. a PHQ-9 score of > 4 (indicative of mild depression);
3. shinkeishitsu-type neurosis including introspective, sensitive, serious, careful, timid, cautious, perfectionistic, or rigid character, assessed by the Diagnostic Interview of Morita shinkeishitsu (DIM);
4. absence of any problems involving injuries, inflammation, or space-occupying lesions at the locations of the acupoints;
5. ability to understand the trial process;
6. no engagement in other forms of activities to improve mood and sleep (e.g., Tai Chi, yoga, and mindfulness meditation) in the last three months before and during the trial.

Exclusion Criteria:

1. severe physical and psychiatric diseases;
2. inability to complete the trial or use necessary psychiatric medicine;
3. cognitive dysfunction caused by neurodegenerative and neurodevelopmental disorders, such as dementia, mental retardation, and autism spectrum disorder;
4. self-injurious or suicidal risk;
5. positive COVID-19 nucleic acid test results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-05-03 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Changes in the Patient Health Questionnaire 9-item depression scale (PHQ-9) | Before and after 2-week treatment immediately.
  The PHQ-9 is a self-report scale which scored each of the DSM-IV diagnostic criteria for major depressive disorders (MDD) from 0 (not at all) to 3 (nearly every day) and total scores of 5, 10, 15, 20 represent mild, moderate, moderately severe, and severe depression, respectively.
Changes in the Generalized Anxiety Disorder 7-item (GAD-7) | Before and after 2-week treatment immediately.
  The GAD-7, comprising seven items scored from 0 to 3 each, is a self-rating scale for generalized anxiety disorder. A total score of 5, 10, or 15 indicated mild, moderate, or severe anxiety symptoms, respectively
Changes in the Insomnia Severity Index (ISI) | Before and after 2-week treatment immediately.
  The ISI could evaluate the severity of current insomnia problems with 7 self-rating items involving staying asleep, falling asleep, waking early morning, noticeability of these problems, distress and daily functioning interference caused by these problems, and sleep satisfaction. A total score ranged from 0 to 28 and cutoff points of 8, 15, and 22 representing subthreshold, moderate, and severe insomnia, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, M.D. Ph.D, Principal Investigator — Central South University
Locations (1):
- Shenzhen Hospital of Integrated Traditional Chinese and Western Medicine, Shenzhen, China